CLINICAL TRIAL: NCT02048267
Title: A Prospective Study of Surgical Outcome and Differences on Histopathology in Patients With Alcoholic & Non Alcoholic Chronic Pancreatitis
Brief Title: Surgical Outcome and Differences on Histopathology in Patients With Alcoholic & Non Alcoholic Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajesh Gupta, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: NK/338/MS/9609-1
Record Dates: First submitted 2014-01-18; First posted 2014-01-29 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Pancreatitis, Chronic
Keywords: Alcoholic; Non alcoholic; Idiopathic; Tropical; Exocrine dysfunction; Endocrine dysfunction; Pain control; Frey's procedure; Duodenum preserving pancreatic head resection
MeSH Terms: conditions — Pancreatitis, Chronic; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Alcoholic
  Interventions: Procedure: Frey's procedure/Pylorus preserving pancreatoduodenectomy
- Non alcoholic
  Interventions: Procedure: Frey's procedure/Pylorus preserving pancreatoduodenectomy

INTERVENTIONS:
Procedure: Frey's procedure/Pylorus preserving pancreatoduodenectomy — Duodenum preserving head resection

SUMMARY:
Numerous treatment modalities have been proposed to treat pain in alcoholic and non-alcoholic chronic pancreatitis such as analgesic medication, inhibition of gastric acid production, enzyme substitution, somatostatin analogues, nerve blockade,reduction of oxidative stress and endoscopic pancreatic duct stenting, but none of these concepts have shown long lasting benefits as surgery in clinical studies.Comparison of surgical outcome in non-alcoholic chronic pancreatitis and alcoholic chronic pancreatitis has limited data and differences on the basis of outcome in between alcoholic and non-alcoholic chronic pancreatitis are not available in literature.

Although it is well known that pain is the main symptom of chronic pancreatitis, it has until now been assessed in very common and varying categories. Pain, however, is only one aspect of the large variety of sensitive facets of daily life. In addition to an improvement in pain symptoms and the preservation of pancreatic exocrine and endocrine function and other parameters, occupational rehabilitation of these mostly young patients and quality of life also should be considered in the evaluation of surgical outcome in alcoholic and non-alcoholic chronic pancreatitis.

In this prospective study, we intend to find out if there are any differences in the surgical outcome on the above mentioned parameters in alcoholic and non-alcoholic chronic pancreatitis.We also plan to see if there are differences in the histopathology in these two disease settings.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of chronic pancreatitis confirmed by at least 2 of the following:

1. Typical Chronic epigastric abdominal pain
2. Elevation of serum Amylase>3 times upper limit normal or
3. Fecal elastase less than 200ug/g stool.
4. Confirmatory findings on cross-sectional imaging:

   1. Changes in size, shape and contour of pancreas
   2. Dilatation of main pancreatic duct
   3. Calcification
   4. Pseudocyst
   5. Pancreatic duct stricture
5. Patients who fulfill the criteria for surgical intervention

Exclusion Criteria:

* Not agreeing for surgical management
* On going acute pancreatitis
* Postop alcohol intake
* Pregnancy.
* Chronic pancreatitis with Malignancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of chronic pancreatitis with unremitting pain requiring surgery at primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | Within first 6 months from the time of surgery
Differences in extent of parenchymal fibrosis, inflammation and ductal obstruction of alcoholic and non alcoholic chronic pancreatitis | Two weeks after surgery

SECONDARY OUTCOMES:
Pain relief | Within first 6 months after surgery
HbA1C,Fasting insulin and C-peptide levels | Within first 6 months after surgery
Fecal elastase levels | Within first 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gupta, M.Ch., Principal Investigator — Professor
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India